CLINICAL TRIAL: NCT06362278
Title: A Multi-omics Study of Patients With Premature Coronary Artery Disease in the Absence of Common Risk Factors
Brief Title: A Multi-omics Study of "Healthy" Premature CAD Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 026
Record Dates: First submitted 2024-01-05; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; multi-omics; premature
MeSH Terms: conditions — Coronary Artery Disease; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 15cc peripheral venous blood will be gathered from each participant for multi-omics studies including: 1）5cc collected with EDTA-K2 tubes for whole-exome study, 2) 5cc collected with PAXGENE tubes for transcriptomics study, 3) 5cc collected with lithium heparin tubes for metabolomics study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cases group: In-patients from cardiology department of The First Affiliated Hospital with Nanjing Medical University will be screened using inclusion/exclusion criteria for patients. Among the patients who meet the criteria and willing to give an informed consent, 30 patients with youngest CAD-diagnosed-age will be enrolled as cases.
  Interventions: Other: multi-omics studies
- matching controls group: In-patients from cardiology department of The First Affiliated Hospital with Nanjing Medical University will be screened using inclusion/exclusion criteria for controls. 30 controls matched in gender and age will be enrolled as matching controls.
  Interventions: Other: multi-omics studies
- verification group: In-patients from cardiology departments of all 3 centers will be screened using inclusion/exclusion criteria. Other than previous 60 participants, about another 100 patients and controls in total who meet the criteria and willing to give an informed consent will be enrolled as verification group.
  Interventions: Other: multi-omics studies

INTERVENTIONS:
Other: multi-omics studies — 15cc peripheral venous blood will be collected for multi-omics studies, including whole-exome study, transcriptomics & metabolomics studies.

SUMMARY:
The goal of this multi-center observational clinical trial is to investigate the genetic risk factors of patients with premature CAD and none traditional CAD risk factors through a multi-omics approach.

The main questions it aims to answer are:

* Genetic risk factors & metabolic fingerprints of patients with premature CAD and none traditional CAD risk factors remain unknown.
* How to optimize current primary prevention strategy for this rare CAD subgroup？

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) remain the leading cause of global mortality despite continuous efforts in disease prevention and treatment optimization. In 2022 alone, CVD caused an estimated 19.8 million deaths worldwide, and ischemic heart disease had the highest global age-standardized DALYs of all diseases at 2,275.9 per 100,000. Therefore, research on the etiology and pathogenesis of coronary artery disease (CAD) remains first priority.

It is now widely known that risk factors such as diabetes mellitus, hyperlipidemia, hypertension, smoking, and obesity are closely related to CAD, but they only explain 30%-40% of CAD risk factors, and large-sample cohort and twin studies have concluded that CAD heritability is estimated to be 40% to 60%. With the development of the Human Genome Project and high-throughput sequencing technology, in the past decade, increasingly larger genome-wide association studies (GWAS) have been conducted worldwide and biobanks established. Public sequencing data is increasingly being used as external common controls instead of sequencing new controls in every study. Till now, thousands of mutations related to CAD have been identified. Multiple Polygenic risk scores (PRSs) have been developed to improve the prediction of common, complex cardiovascular diseases like CAD on individual level.

Premature CAD has been proved to have strong link with family history of cardiovascular and cerebral vascular disease, which indicates a strong genetic background of premature CAD. However, there is an even more scarce & inconspicuous subgroup of premature CAD, defined as premature CAD without common CAD risk factors in this study. First of all, most of those patients were considered "healthy" or "at very low risk of CVDs" before CAD was diagnosed; secondly, genetic risk factors & metabolic fingerprints of such patients remain unknown; thirdly, we still don't know yet how to optimize current primary prevention strategy for this rare CAD subgroup.

For this regard, we designed this multi-omics study to cover the questions mentioned above.

ELIGIBILITY:
Inclusion Criteria for cases:

1. In-patients from cardiology department of either following 3 hospitals: a) The First Affiliated Hospital of Nanjing Medical University; b) Qilu Hospital of Shandong University; c) The Second Affiliated Hospital Zhejiang University School of Medicine
2. Confirmed diagnosis of Obstructive CAD (≥50% diameter stenosis in a major epicardial vessel) through coronary angiography
3. Age of the patient when Obstructive CAD was for the first time diagnosed should be no more than 45 years old for the male and 55 years old for the female.

Inclusion Criteria for controls:

1. In-patients from cardiology department of either following 3 hospitals: a) The First Affiliated Hospital of Nanjing Medical University; b) Qilu Hospital of Shandong University; c) The Second Affiliated Hospital Zhejiang University School of Medicine
2. Coronary artery stenosis was ruled out through either coronary angiography or coronary CTA.

Exclusion Criteria for both cases and controls:

1. Patients with hypertension (grade 1-3)
2. Patients with type 1 or type 2 diabetes mellitus
3. BMI >28.0 Kg/m^2
4. Patients with non-ideal blood lipids level on admission(defined as either LDL-C≥2.6mmol/L OR non-HDL cholesterol≥3.4mmol/L OR Lipoprotein(a) ≥300mg/L)
5. Smoker (Smoking for more than 6 consecutive or cumulative months in a lifetime, whether quit smoking or not)
6. Patients with hyperuricemia or gout
7. eGFR<60 ml/min·1.73m^2
8. Patients with structural heart diseases, inherited cardiomyopathies & arrhythmias
9. Other reasons a participant considered unsuitable for inclusion by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In-patients from cardiology department of either following 3 hospitals: a) The First Affiliated Hospital of Nanjing Medical University; b) Qilu Hospital of Shandong University; c) The Second Affiliated Hospital Zhejiang University School of Medicine. Those patients who meet the criteria for cases or controls and willing to give an informed consent will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
common & rare variants associated with "healthy" pre-mature CAD phenotype | 3 months
  Whole-exome study in both patients and matching controls will be pefromed using rare-variant collapsing analyses to findout common & rare variants accosicated with this phenotype. Relative variants will be further screend & validated in verification group. If necessary, further casade screening using trios-wes technique will be perfromed within certain families under written consent.
Unique metabolomic fingerprints associated with "healthy" pre-mature CAD phenotype | 3 months
  Non-targeted metabonomic analysis of plasma will be performed in both patients and matching controls. Relative metabolites will be further screend & validated in verification group. If necessary, further targeted metabonomic analysis will be performed using redundant serum samples .

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (3):
- China (3):
  - First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Qilu Hospital of Shangdong University, Jinan, Shandong
  - The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be published until further permission granted from domestic Human Genetic Resource Administration.

REFERENCES:
- [Background] Mensah GA, Fuster V, Murray CJL, Roth GA; Global Burden of Cardiovascular Diseases and Risks Collaborators. Global Burden of Cardiovascular Diseases and Risks, 1990-2022. J Am Coll Cardiol. 2023 Dec 19;82(25):2350-2473. doi: 10.1016/j.jacc.2023.11.007. No abstract available. PMID 38092509
- [Background] Kessler T, Vilne B, Schunkert H. The impact of genome-wide association studies on the pathophysiology and therapy of cardiovascular disease. EMBO Mol Med. 2016 Jul 1;8(7):688-701. doi: 10.15252/emmm.201506174. Print 2016 Jul. PMID 27189168
- [Background] O'Sullivan JW, Raghavan S, Marquez-Luna C, Luzum JA, Damrauer SM, Ashley EA, O'Donnell CJ, Willer CJ, Natarajan P; American Heart Association Council on Genomic and Precision Medicine; Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Lifestyle and Cardiometabolic Health; and Council on Peripheral Vascular Disease. Polygenic Risk Scores for Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2022 Aug 23;146(8):e93-e118. doi: 10.1161/CIR.0000000000001077. Epub 2022 Jul 18. PMID 35862132
- [Background] Muse ED, Chen SF, Torkamani A. Monogenic and Polygenic Models of Coronary Artery Disease. Curr Cardiol Rep. 2021 Jul 1;23(8):107. doi: 10.1007/s11886-021-01540-0. PMID 34196841
- [Background] Saadatagah S, Varughese MG, Nambi V. Coronary Artery Disease Risk Prediction in Young Adults: How Can We Overcome the Dominant Effect of Age? Curr Atheroscler Rep. 2023 Jun;25(6):257-265. doi: 10.1007/s11883-023-01106-1. Epub 2023 May 17. PMID 37195598
- [Background] Vilne B, Schunkert H. Integrating Genes Affecting Coronary Artery Disease in Functional Networks by Multi-OMICs Approach. Front Cardiovasc Med. 2018 Jul 17;5:89. doi: 10.3389/fcvm.2018.00089. eCollection 2018. PMID 30065929
- [Background] Collet JP, Zeitouni M, Procopi N, Hulot JS, Silvain J, Kerneis M, Thomas D, Lattuca B, Barthelemy O, Lavie-Badie Y, Esteve JB, Payot L, Brugier D, Lopes I, Diallo A, Vicaut E, Montalescot G; ACTION Study Group. Long-Term Evolution of Premature Coronary Artery Disease. J Am Coll Cardiol. 2019 Oct 15;74(15):1868-1878. doi: 10.1016/j.jacc.2019.08.1002. PMID 31601367
- [Background] Navas-Nacher EL, Colangelo L, Beam C, Greenland P. Risk factors for coronary heart disease in men 18 to 39 years of age. Ann Intern Med. 2001 Mar 20;134(6):433-9. doi: 10.7326/0003-4819-134-6-200103200-00007. PMID 11255518
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Singh A, Collins BL, Gupta A, Fatima A, Qamar A, Biery D, Baez J, Cawley M, Klein J, Hainer J, Plutzky J, Cannon CP, Nasir K, Di Carli MF, Bhatt DL, Blankstein R. Cardiovascular Risk and Statin Eligibility of Young Adults After an MI: Partners YOUNG-MI Registry. J Am Coll Cardiol. 2018 Jan 23;71(3):292-302. doi: 10.1016/j.jacc.2017.11.007. Epub 2017 Nov 12. PMID 29141201
- [Background] Wojcik GL, Murphy J, Edelson JL, Gignoux CR, Ioannidis AG, Manning A, Rivas MA, Buyske S, Hendricks AE. Opportunities and challenges for the use of common controls in sequencing studies. Nat Rev Genet. 2022 Nov;23(11):665-679. doi: 10.1038/s41576-022-00487-4. Epub 2022 May 17. PMID 35581355